CLINICAL TRIAL: NCT00129285
Title: A Double-Blind, Placebo-Controlled Study of Modafinil for Cocaine Dependence
Brief Title: Modafinil Treatment for Cocaine-Dependent Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-15366-1; R01DA015366 (NIH); DPMC (Other: NIDA); 704450
Record Dates: First submitted 2005-08-04; First posted 2005-08-11 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose Modafinil (Experimental): Low Dose Modafinil 200 mg daily
  Interventions: Drug: Low Dose Modafinil
- High Dose Modafinil (Experimental): High dose modafinil 400 mg daily
  Interventions: Drug: High Dose Modafinil
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose Modafinil — modafinil 200 mg/day
  Other Names: Provigil
  Arms: Low Dose Modafinil
Drug: High Dose Modafinil — modafinil 400 mg/day
  Other Names: Provigil
  Arms: High Dose Modafinil
Drug: Placebo — placebo 400 mg/day
  Arms: Placebo

SUMMARY:
Despite years of active research, there are still no approved medications for the treatment of cocaine dependence. The purpose of this study is to determine the effectiveness of modafinil in treating cocaine-dependent individuals.

DETAILED DESCRIPTION:
Modafinil is a glutamate-enhancing agent that blunts cocaine euphoria under controlled conditions. Due to its stimulant-like properties, modafinil is also likely to relieve severe cocaine withdrawal symptoms. In turn, this may lead to better clinical outcomes. The purpose of this study is to determine whether modafinil improves abstinence during early recovery from cocaine dependence.

This 6-month, double-blind, placebo-controlled trial will enroll 210 participants with current DSM-IV diagnoses of cocaine dependence. Treatment will occur for 8 weeks. Participants will be randomly assigned to receive a single morning dose of low-dose modafinil (200 mg/day), high-dose modafinil (400 mg/day), or matching placebo tablets. In addition, each week participants will receive manual-guided cognitive behavioral therapy at the Treatment Research Center. At the end of the 8-week treatment period, modafinil or placebo will be abruptly discontinued. One week following, an end of medication evaluation will occur. In addition to this, two follow-up evaluations will take place 3 and 5 months after initial randomization. Efforts will be made to continue evaluation of subjects who decide to discontinue the modafinil treatment. Urine benzoylecgonine levels will be used to measure cocaine abstinence. Craving, withdrawal, retention, and adverse events will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 - 60 years;
* Current DSM-IV diagnosis of cocaine dependence
* Using at least $200 worth of cocaine within the past 30 days and having positive urine toxicology (BE) during screening;
* Able to provide written informed consent and to comply with all study procedures;
* Women must be surgically sterile, at least two years postmenopausal, or if of childbearing potential be using a medically accepted method of birth control and agree to continue use of this method for at least 30 days after the last dose of study drug (i.e. barrier method with spermicide, steroidal contraceptive [oral and implanted, including Depo-Provera contraceptives must be used in conjunction with a barrier method], or intrauterine device [IUD])

Exclusion Criteria:

* Currently dependent on any substance other than cocaine or nicotine
* Neurological or psychiatric disorders, such as psychosis, bipolar illness, organic brain disease, dementia, or any diseases that require psychotropic medications
* Serious medical illnesses, including but not limited to; uncontrolled hypertension, significant heart disease (including a history of myocardial infarction, angina, mitral valve prolapse, left ventricular hypertrophy, palpitations, and arrhythmia), hepatic disease, renal disease, or any serious, potentially life-threatening or progressive medical illness that may compromise patient safety or study conduct;
* Received a drug with known potential for toxicity to a major organ system within the month prior to entering treatment including but not limited to; chemotherapeutic agents for neoplastic disease (i.e. methotrexate, vincristine, vinblastine, fluorouracil), agents used for parasitic infections, isoniazid, chlorambucil, dactinomycin, chloramphenicol, immunosuppressive and cytotoxic agents (i.e. cyclosporine, tacrolimus), indomethacin, protease inhibitors, amphotericin B, cephalosporins, aminoglycosides, interferon, and sulfonamides;
* Clinically significant abnormal laboratory values
* Has any disease of the gastrointestinal system, liver, or kidneys which could result in altered metabolism or excretion of the study medication (history of major gastrointestinal tract surgery, gastrectomy, gastrostomy, bowel resection, etc.) or history of chronic gastrointestinal disorders (ulcerative colitis, regional enteritis, or gastrointestinal bleeding);
* Known hypersensitivity or allergy to modafinil or receiving chronic therapy with any medication that could interact adversely with one of the medications under study, including propranolol, phenytoin, warfarin and diazepam;
* Currently taking any medication that could interact adversely with one of the medications under study, including propranolol, phenytoin, warfarin and diazepam
* Took monoamine oxidase inhibitors (MAOI) within 30 days prior to randomization;
* Taking or has taken an investigational drug within 60 days prior to enrollment
* If female and of child-bearing capacity, tests positive on a urine pregnancy test, is lactating, has had three or more days of amenorrhea beyond expected menses at the time of the first dose of study medication, is contemplating pregnancy in the next 6 months, or is not using an effective contraceptive method;
* Received therapy with any opiate-substitute (methadone, LAAM, buprenorphine) within 60 days of study enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2004-07; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Dackis, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Click here for more information about the University of Pennsylvania Treatment Research Center's current studies — http://www.med.upenn.edu/csa/trc_clinical_trials.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Modafinil: Low Dose Modafinil
  Modafinil Low Dose: participants received modafinil 200 mg/day
- High Dose Modafinil: High Dose Modafinil
  Modafinil High Dose: participants received modafinil 400 mg/day
- Placebo: Placebo
  Placebo: participants received placebo 400 mg/day
Period: Overall Study
Arm/Group | Low Dose Modafinil | High Dose Modafinil | Placebo
Started | 65 | 70 | 75
Completed | 40 | 43 | 37
Not Completed | 25 | 27 | 38

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Modafinil: Low Dose Modafinil
  Modafinil Low Dose: modafinil 200 mg/day
- High Dose Modafinil: High Dose Modafinil
  Modafinil High Dose: modafinil 400 mg/day
- Total: Total of all reporting groups
Arm/Group | Low Dose Modafinil | High Dose Modafinil | Placebo | Total
Number analyzed (Participants) | 65 | 70 | 75 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 65 | 70 | 75 | 210
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.72 (6.9) | 43.64 (7.7) | 42.46 (7.5) | 42.64 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 19 | 55
  Male | 47 | 52 | 56 | 155
Region of Enrollment [Number; unit: participants]
  United States | 65 | 70 | 75 | 210

OUTCOME MEASURES:

1. Primary Outcome: Urine Toxicology for Cocaine
Description: Abstinent in the final 3 weeks of treatment
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Modafinil | High Dose Modafinil | Placebo
Number analyzed (Participants) | 65 | 70 | 75
Participants | 3 | 8 | 3

2. Secondary Outcome: Retention; Number of Evaluation Visits Attended
Description: Number of visits attended compared between the three conditions using anova
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: number of evaluation sessions attended
Groups:
- 1Low Dose Modafinil: Low Dose Modafinil 200 mg daily
  Modafinil Low Dose: modafinil 200 mg/day
- 2 High Dose Modafinil: High Dose Modafinil 400 mg daily
  Modafinil High Dose: modafinil 400 mg/day
- 3. Placebo: Placebo
  Placebo: placebo 400 mg/day
Arm/Group | 1Low Dose Modafinil | 2 High Dose Modafinil | 3. Placebo
Number analyzed (Participants) | 65 | 70 | 75
number of evaluation sessions attended | 16.8 (7.1) | 16.5 (6.7) | 14.3 (7.1)

3. Secondary Outcome: Cocaine Selective Severity Assessment (CSSA) Total Score
Description: Cocaine Selective Severity assessment (CSSA) total score has a range 0-126. Higher scores indicating greater severity of cocaine withdrawal obtained weekly. Groups compared using GEE model over 8 weeks of treatment.
Time Frame: 8 weeks
Population: patients exposed to low dose and high dose modafinil
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: received placebo
Arm/Group | Low Dose Modafinil | High Dose Modafinil | Placebo
Number analyzed (Participants) | 65 | 70 | 75
units on a scale | 12.89 (11.70) | 15.04 (13.52) | 15.2 (14.32)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of the 8 week trial
Description: Adverse events for low and high dose modafinil were combined and compared to adverse events occurring in the placebo comparator group.
Groups:
- Modafinil High Dose: Modafinil 400 mg daily
- Placebo: Placebo daily
- Modafinil Low Dose: modafinil 200 mg daily
Arm/Group | Modafinil High Dose | Placebo | Modafinil Low Dose
Serious Adverse Events (participants affected / at risk) | 1/70 | 0/75 | 0/65
Other Adverse Events (participants affected / at risk) | 63/70 | 62/75 | 50/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil High Dose (N=70) | Placebo (N=75) | Modafinil Low Dose (N=65)
Treatment Emergent Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Modafinil High Dose (N=70) | Placebo (N=75) | Modafinil Low Dose (N=65)
Headache (General disorders) | 15 | 14 | 11
Body Aches (Musculoskeletal and connective tissue disorders) | 23 | 27 | 17
Upper respiratory tract infection (Infections and infestations) | 18 | 22 | 14
Insomnia (General disorders) | 9 | 5 | 6
teeth problems (General disorders) | 6 | 7 | 6
Increased energy (Nervous system disorders) | 10 | 2 | 6
appetite changes (Gastrointestinal disorders) | 4 | 8 | 6
Nausea (Gastrointestinal disorders) | 4 | 4 | 5
Diarrhea (Gastrointestinal disorders) | 6 | 4 | 2
Stomach problems (Gastrointestinal disorders) | 6 | 4 | 2
Dry mouth (General disorders) | 3 | 3 | 5
Fatigue (General disorders) | 4 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No